CLINICAL TRIAL: NCT03421262
Title: Pregnancy Outcomes and Medical Costs According to Gestational Diabetes Mellitus Diagnostic Criteria: Randomized Prospective Study.
Brief Title: Pregnancy Outcomes and Medical Costs According to Gestational Diabetes Mellitus Diagnostic Criteria
Acronym: POMEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00003
Record Dates: First submitted 2017-11-27; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-step:IADPSG Criteria (Experimental): Gestational diabetes screening with fasting 2 hour 75g. Receive a fasting 2 hour 75 gr oral glucose tolerance test and diagnosed based on the IADPSG which is if one or more values exceed the following diagnostic threshold: Fasting 92, 1-hour 180, or 2-hour 153 mg/dL.
  Interventions: Diagnostic Test: IADPSG Criteria
- Two-step:NDDG Criteria (Active Comparator): Step 1: Perform a 1h 50-g glucose load test (nonfasting. If the plasma glucose level measured 1 h after the load is 140 mg/dL, proceed to a 100-g OGTT.
  Step 2: 100-g OGTT. The diagnosis of GDM is made if at least two of the following four plasma glucose levels(measured fasting and 1 h, 2 h, 3 h after the OGTT) are met or exceeded: 105mg/dl, 190mg/dl, 165mg/dl and 145mg/dl respectively
  Interventions: Diagnostic Test: NDDG Criteria

INTERVENTIONS:
Diagnostic Test: IADPSG Criteria — One-step: 2 hr 75 gr OGTT
  Arms: One-step:IADPSG Criteria
Diagnostic Test: NDDG Criteria — Osullivan test + 3 h 100 g OGTT
  Arms: Two-step:NDDG Criteria

SUMMARY:
The aim of the study is to evaluate differences in pregnancy outcomes and medical costs depending on gestational diabetes diagnostic criteria used (one vs two-step approach).

DETAILED DESCRIPTION:
Due to Hyperglycemia and Adverse Pregnancy Outcomes study results, a new gestational diabetes mellitus (GDM) diagnostic criteria was defined using a one-step approach (75-g oral glucose tolerance test -OGTT-).

However, not all scientific societies have accepted and have implanted this new diagnostic criteria. The lowest glycemia cut-off of this criteria regarding the two-step approach entails an increase in GDM incidence with discordant studies about its cost-effectivity.

It will be assessed if pregnancy outcomes and medical costs are different depending on diagnostic criteria used.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* No expectation that subject will be moving out of the area of the clinical center during the next year
* Informed Consent Form signed by the subject

Exclusion Criteria:

* Preexisting type 1 or 2 diabetes
* Advanced HIV( on medications that cause hyperglycemia), severe liver disease, gastric bypass surgery or other illness/surgeries that preclude them from drinking the glucose solution.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3644 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-27 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Large for gestational age | At birth of infant
  Infant birthweight >90th centile using customized growth curves

SECONDARY OUTCOMES:
Macrosomia | At birth of infant
  infant birthweight >=4kg
Small for gestational age | At birth of infant
  infant birthweight <10th centile using customized growth curves
Hypertension in pregnant | First 3 months postpartum
  classification according to American College of Obstetricians and Gynecologists (Task Force on Hypertension in Pregnancy).
Neonatal obstetric trauma | At birth of infant
  rate of shoulder dystocia, clavicle fracture, brachial plexus injury and intrapartum asphyxia
Congenital anomalies | At birth of infant
  Coding of EUROCAT
Neonatal hypoglycemia | up to 4 weeks after delivery
  neonatal plasma glucose levels of <2.5 mmol/L in the first 24 hours of life and <2.8 mmol/L thereafter.
Neonatal hypocalcemia | up to 4 weeks after delivery
  neonatal calcium levels of <7mg/dl
Neonatal hyperbilirubinemia | up to 4 weeks after delivery
  hyperbilirubinemia treated with phototherapy
Neonatal polycythemia | up to 4 weeks after delivery
  hematocrit from a peripheral venous sample is >65 percent
Respiratory Distress Syndrome | up to 4 weeks after delivery
  onset of progressive respiratory failure shortly after birth, in conjunction with a characteristic chest radiograph (after ruling out other causes).
Infant Outcomes | up to 4 weeks after delivery
  Pregnancy loss (Miscarriage, stillbirth, neonatal death)
Hypertrophic cardiomyopathy | up to 4 weeks after delivery
  increased left ventricular (LV) wall thickness ≥15 mm is imaged anywhere in the LV wall (by transthoracic echocardiography)
Polyhydramnios | At birth of infant
  Amniotic fluid index ≥25 cm
Gestational age at delivery | At birth of infant
  Gestational age was defined as completed weeks based on last menstrual period or the earliest ultrasound assessment if discordant.
Cesarean section | At birth of infant
  delivery of a baby through a surgical incision in the mother's abdomen and uterus
Perinatal mortality | First 7days postpartum
  infant deaths that occur at less than 7 days of age and fetal deaths with a gestational age of 28 weeks or more.
NICU admission | up to 4 weeks after delivery
  NICU admission for treatment or surveillance
Maternal hospital stay | up to 4 weeks from maternal discharge
  Length of hospital stay (days)
Neonatal hospital stay | up to 4 weeks from neonatal discharge
  Length of hospital stay (days)
Evaluation of mediterranean diet adherence | up to 12-14weeks from last menstrual period.
  using Mediterranean Diet Adherence Screener (MEDAS) questionnaire. Score betwwen 0-14; high score indicate maximum mediterranean diet adherence.
Evaluation of health-related physical activity | up to 12-14weeks from last menstrual period.
  using International Physical Activity Questionnaire (IPAQ). Data collected with IPAQ can be used as a continuous measure (Metabolic Equivalent of Task [MET]-minutes/week) or caterorical measure (low, moderate or high physical activity)
Medical cost | First 3 months postpartum
  Economic cost include: laboratory costs; glucose bottles (50 g, 100 g and 75 g); pharmaceutical expenditure (exact insulin doses consumed, total pens, needles, strips); medical visits during pregnany and postpartum (endocrinologist,educational nurses, obstetrician and midwifes); total number of tests (ultrasonds, cardiotocography record); cost of intensive care unit admissions (Length of stay and complexity) and total hospital admission costs.
  All these variables will be expressed as cost (€).

CONTACTS AND LOCATIONS:
Overall Officials: Verónica Perea, MD, Principal Investigator — Hospital Universitari Mutua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03421262/Prot_SAP_000.pdf